CLINICAL TRIAL: NCT02148458
Title: Metabolic and Molecular Effects of a Mediterranean Diet and Intermittent Fasting
Brief Title: Short Term Intermittent Fasting and Mediterranean Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201404045
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Overweight; Pre-hypertension; Hypertension; Hypercholesterolemia; Glucose Intolerance
Keywords: Intermittent fasting; Mediterranean diet; overweight; Calorie restriction
MeSH Terms: conditions — Overweight; Prehypertension; Hypertension; Hypercholesterolemia; Glucose Intolerance; Intermittent Fasting | interventions — Diet, Mediterranean; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): Western diet for 8 weeks, followed by 8 weeks of Western diet with intermittent fasting.
  Interventions: Other: Control group
- Mediterranean diet (Experimental): Mediterranean diet for 8 weeks, followed by 8 weeks of Mediterranean diet with intermittent fasting.
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Other: Mediterranean diet — Mediterranean diet for 8 weeks, followed by 8 weeks of Mediterranean diet with intermittent fasting (i.e. 2 non-consecutive days of fasting per week)
  Arms: Mediterranean diet
Other: Control group — control group eating their usual Western diet for 8 weeks, followed by 8 weeks of usual diet with intermittent fasting (i.e. 2 non-consecutive days of fasting per week).
  Arms: Control group

SUMMARY:
The purpose of this research study is to evaluate the effects of intermittent fasting in subjects that are eating a Mediterranean diet or a Western diet. This study is part of ongoing research in the prevention and treatment of age-related diseases at Washington University School of Medicine.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether or not IF, independently of changes in quality of diet, reduces the level of chronic inflammation as evidenced by a decrease in high sensitivity C-reactive protein (hsCRP), as the main outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. - The participants in this study will be 50 men and women in the 30 to 65 year age range, who have a BMI in the high-normal to moderately overweight range (i.e. 22 to 28 kg/m2),
2. - Participants who are eating usual US diets and are sedentary to moderately active (i.e. not exercise trained).
3. - Participants have at least one of these metabolic abnormalities: pre-hypertension or hypertension (i.e. systolic blood pressure > 120 mmHg or diastolic blood pressure > 80 mmHg or specific treatment of previously diagnosed hypertension)10, sub-optimal lipid levels (i.e. LDL-cholesterol > 100 mg/dl or HDL-cholesterol < 59 mg/dl or specific treatment for this lipid abnormality)11, impaired fasting glucose or glucose intolerance (i.e. fasting glucose > 100 mg/dl or 2 hr-glucose during OGTT with a glucose load of 75 g > 140 mg/dl or specific treatment for previously diagnosed type 2 diabetes)12, or high-risk waist circumference (≥ 94 cm in men and ≥ 80 cm in women)13.

Exclusion Criteria:

- 1 - History of any chronic disease process that could interfere with interpretation of results 2 - Smoking, pregnancy, alcoholism, psychiatric problems, life situations that would interfere with study participation and compliance.

3 - Currently eating diet similar to Mediterranean diet based on dietary and food frequency questionnaires and 4-day food diary.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Decrease in high sensitivity C-reactive protein (hsCRP) | 16 weeks-- Baseline, 8 weeks, 16 weeks
  hsCRP is in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Tosti, MD, Principal Investigator — Washington University School of Medicine; Luigi Fontana, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University school of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Plan to publish

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717